CLINICAL TRIAL: NCT05017740
Title: A Randomised Clinical Trial in the Use of Physiological Intra-cytoplasmic Spermatozoa Injection (PICSI) in Couples With a Previous Poor Fertilisation Cycle in In-vitro Fertilisation.
Brief Title: PICSI RCT in Couples With a Previous Poor Fertilisation Cycle in IVF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/RM/001
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Infertility; IVF
Keywords: PICSI
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to undergo PICSI or standard ICSI in a 1:1 treatment ratio.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Trial participants, research team collecting data outcome, and all study team members except the embryologists will be blinded to treatment allocation. It is not possible to conceal allocation to the embryologists, who will perform the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI (Active Comparator)
  Interventions: Procedure: ICSI
- PICSI (Active Comparator)
  Interventions: Procedure: PICSI

INTERVENTIONS:
Procedure: ICSI — In ICSI, the sperm is chosen based on motility and gross morphology to be inseminated directly into the cytoplasm of the oocyte.
  Arms: ICSI
Procedure: PICSI — In PICSI, the sperm is selected via hyaluronic binding before insemination into the cytoplasm of the oocyte.
  Arms: PICSI

SUMMARY:
Poor fertilisation plays a significant role in poor artificial reproductive technique outcomes. Male factor infertility accounts for a large portion of such cases. Several modalities have been proposed as a solution, including physiological intra-cytoplasmic sperm injection (PICSI). PICSI is a technique used to select the sperm to use in intra-cytoplasmic sperm injection (ICSI) treatment. It involves placing sperm with hyaluronic acid, a natural compound found in the body. PICSI identifies sperm that can bind to hyaluronic acid and these sperms are selected for use in treatment.

Some studies have suggested that PISCI may be advantageous to reduce miscarriage. However, the evidence is not strong and it remains unknown if PICSI is effective in a selected group of couples with a history of poor fertilisation. Based on previous medical records, we observed a higher clinical pregnancy rate (CPR) and a trend towards lower miscarriage rates with PICSI. To verify the findings and address the clinical gap, we propose a randomised controlled trial (RCT) with 234 couples (117 in each group) to evaluate the effectiveness of PICSI comparing with ICSI for improving CPR and reducing miscarriage rate in couples with a fertilisation rate of <50% in their first cycle of ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Couples with <50% fertilisation in their first ICSI cycle, and scheduled for their second ICSI/PICSI cycle

Exclusion Criteria:

* Women with diminished ovarian reserves (AMH <1.2ng/ml) or severe endometriosis (rAFS Stage III or IV)
* Male partner with severe oligoasthenoteratozoospermia (Density < 5 million, Total motility < 40) or those require surgically retrieved sperm
* Couples using donor gametes
* Couples using frozen gametes
* Couples undergoing split IVF-ICSI cycles
* Couples where a freeze all approach has been done, either clinically indicated or secondary to patient choice

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6-9 weeks after fresh embryo transfer
  The presence of fetal heartbeat or gestational sac at 6-9 weeks after fresh embryo transfer
Miscarriage rate | 6 to 23+6 gestational weeks
  Pregnancy loss before 23+6 completed weeks after confirmation of clinical pregnancy

SECONDARY OUTCOMES:
Fertilisation rate | 2-5 days after oocyte retrieval
  Successful embryo transfer
Live birth rate | After 24 completed weeks of gestation
  Live birth after 24 completed weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Chan, MB BCh BaO MA FRCOG PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No